CLINICAL TRIAL: NCT04163133
Title: Comparison of Regular Trigger Timing and 1～2 Days Delay of Trigger in Ovarian Stimulations by GnRH Antagonist Protocol in in Vitro Fertilization
Brief Title: Trigger Timing in Ovarian Stimulations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Li Rong, Director of Reproductive Medical Center, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2019261
Record Dates: First submitted 2019-11-06; First posted 2019-11-14 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: IVF Outcome
Keywords: delay of trigger, ovarian stimulation, antagonist protocol

STUDY DESIGN:
Intervention Model Description: A single center, open-label, randomized controlled clinical trial (1:1 treatment ratio). On the day of regular trigger timing day (three follicles reach 17mm) or 1～2 days later. 36(±2) hours after trigger, oocyte retrieval will be applying in both group with same protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1～2 days delay of trigger group (Experimental): 1～2 days later of trigger than regular trigger timing day (three follicles reach 17mm) .
  Interventions: Procedure: 1～2 days later trigger than regular timing
- regular trigger group (No Intervention): regular trigger timing when three follicles reach 17mm bilateral.

INTERVENTIONS:
Procedure: 1～2 days later trigger than regular timing — During ovarian stimulation, 1～2 days later of trigger after three follicles reach 17mm bilateral with contineous using of Gonadotrophin in antagonist protocol.
  Arms: 1～2 days delay of trigger group

SUMMARY:
The use of antagonist ovulation stimulation program is increasing year by year, because of its convenience, flexibility, and prevention effect of ovarian hyperstimulation syndrome. However, many researchers and clinicians believe that the clinical outcomes of antagonist regimens are worse than those of classical long-term regimens. Studies showed that the reasons for that maybe antagonist protocol results in poor effect on oocytes maturation or endometrial receptivity.

At present, the trigger time of antagonist regimen is more than three follicles with diameters of ≥17 mm, which makes the duration of gonadotrophin application in antagonist regimen is shorter than that of long regimen. Whether the trigger time of antagonist regimen is too early to cause adverse effects on oocytes, embryos and eventual clinical outcomes is unknown.

This study hopes to compare regular trigger timing and 1～2 days delay of trigger in ovarian stimulations by antagonist protocol，in order to study whether delay 1～2 days of trigger will get better clinical outcomes than regular trigger timing in ovarian stimulations by antagonist protocol in in vitro fertilization (IVF)/Intracytoplasmic sperm injection (ICSI).

The results of this study will help infertile couples and clinicians to know and choose the optimal treatment in antagonist protocol.

DETAILED DESCRIPTION:
The objective of this study is to conduct a single center clinical trial, to study whether delay 1～2 days of trigger will obtain more good-quality embryos than regular trigger timing in ovarian stimulations by antagonist protocol in in vitro fertilization. Which may further improve culmulative live birth rate (CLBR). The results of this study will help infertile couples and clinicians to know and choose the optimal treatment in antagonist protocol.

We plan a single center, open-label, randomized controlled clinical trial (1:1 treatment ratio). On the day of regular trigger timing day (three follicles reach 17mm) or 1～2 days later. 36-38 hours after trigger, oocyte retrieval will be applying in both group with same protocol. Then IVF/ICSI and embryo culture with standard protocol in assisted reproductive treatments in our center will be implemented similarly. Information of all participants and outcomes are recorded in the case report form. The flow chart followed SPIRIT checklist showing enrollment, allocation, treatment, and follow-up of participants.

Inclusion Criteria:

* Age: ≥18 and <42 years old
* Antral follicle count (AFC): ≥5 and <20
* Anti-mullerian hormone (AMH): ≥1.1 ng/mL and <2.5 ng/mL
* Body mass index (BMI): ≥18.5 Kg/m2 and <29 Kg/m
* First or second ART cycle
* Regular menstrual cycles (between 22 and 35 days)
* Two ovaries present
* Planned for single or double day 3 transfer
* Infertile couples scheduled for their first IVF/ICSI cycle with fixed antagonist protocol.
* Informed consent obtained.

Exclusion criteria:

* Women with contraindication for IVF or ICSI, such as poorly controlled type 1 or type 2 diabetes mellitus; undiagnosed liver disease or dysfunction (based on serum liver enzyme test results); renal disease or abnormal serum renal function; significant anemia; history of deep venous thrombosis, pulmonary embolus or cerebrovascular accident; uncontrolled hypertension or known symptomatic heart disease; history of (or suspected) cervical carcinoma, endometrial carcinoma or breast carcinoma; and undiagnosed vaginal bleeding.
* Previous history of poor ovarian response (<4 oocytes retrieved) with a maximal dose of ovarian stimulation (OS) (≥300 IU/day) or ovarian hyperstimulation syndrome (OHSS), regardless of gonadotropin dose
* Known reasons for impaired implantation (i.e. hydrosalpinx, fibroid distorting the endometrial cavity, Asherman's syndrome, thrombophilia or endometrial tuberculosis)
* Repeated miscarriages (>2 previous biochemical pregnancies or >2 spontaneous miscarriages)
* Recurrent implantation failure (>3 failed cycles with good quality embryos)
* Polycystic ovary syndrome (PCOS)
* Untreated thyroid disfunction
* Administration of exogenous E2, P4 or gonadotropins in the preceding menstrual cycle
* Active female smoking
* Ongoing pregnancy
* Women who have previously enrolled in the trial
* Those unable to comprehend the investigational nature of the proposed study
* either male partner or female partner has to receive donor sperm or donor eggs.
* Either male partner or female partner has to receive preimplantation genetic diagnosis (PGD) and preimplantation genetic screening (PGS).

Withdrawal criteria:

* Participants who are unwilling to continue the trial procedures or withdraw the informed consent.
* Participants who appear poor compliance during the trial, and researchers confirm it is necessary to discontinue their study.
* Loss to follow-up. Recruitment Infertile couples who come to outpatient clinic will be screened as part of routine assessment by trained clinical team who are very familiar with the eligible criteria. Eligible patients will then be approached by a member of the research team and explained the trial details before controlled ovarian hyperstimulation (COH). After this information, couples will be offered time for consideration to decide to participate the trial. If the couple agrees to participate, they will make an appointment to sign the consent before COH. Couples that refuse participation, will receive conventional care. An individual record of all non-recruited patients and reasons for exclusion will be obtained and storage.

Controlled ovarian hyperstimulation All patients will receive fixed antagonist protocol of COH treatment, which is performed by standard routines at each study center. Treatment will start on day 2 or day 3 of the spontaneous menstrual cycle, and the baseline pelvic ultrasound, as well as basic serum hormones (such as FSH, luteinizing hormone (LH), progesterone (P) and β-hCG) will be tested to confirm the folic status. All participants will be subcutaneous injected rFSH. The initial dosage of rFSH is 200IU and the subsequent dose will be adjusted according to the ovary status. Transvaginal B-mode ultrasound, urinary LH, and serum E2 will be tested to monitor follicle growth. On day 5 of stimulation, GnRH antagonist 0.25mg daily will be administered subcutaneously until the trigger day (include the trigger day). Group A of trigger is 3 or more follicles reach a diameter ≥17 mm, Group B of trigger is 1～2 days later than group A with continually Gn.

Oocyte retrieval and preparation Oocyte retrieval is scheduled for 36h (±2) after hCG injection. Routine oocyte pick-up is performed under Transvaginal ultrasound guidance via 17G oocyte aspiration needle with use of intravenous sedation. The retrieved cumulus oocyte complexes (COC) will be allocated to undergo conventional IVF or ICSI. For both groups, the COCs are placed in culture medium covered by lightweight paraffin oil and incubated in a humidified 37℃,5% CO2 incubator after oocyte retrieval immediately. Besides of this, the COCs are incubated for 2-6h before insemination or injection. For group B (ICSI group), the oocytes will be denuded by hyaluronidase before micromanipulation. Only the mature, metaphase-Ⅱ(MⅡ) oocytes with an extruded first polar body are microinjected.

Assessment of fertilization and embryo quality Assessment of fertilization are carried out about 16-18h (day 1) after fertilization. Oocytes are classed as fertilized if two pronuclei (2PN) are present and the second polar body has been extruded. Other oocytes are classified as abnormally fertilized (0PN, 1PN, 3PN). Normal fertilization rate will be always calculated as the number 2PN over the number of COCs, independent of the nuclear maturity, as well for IVF as for ICSI. After the evaluation on day 1, zygotes are left in culture for a further 48 hours, and the cleavage embryo quality will be observed at 72 (day 3) hours after oocyte retrieval. The embryos are scored according to the quality, numbers, size of the blastomeres and the amount of anucleate fragmentation as follow criteria: Grade 1 embryos consist of symmetrical blastomeres of approximately equal size and without anucleate fragments. Grade 2 embryos had blastomeres of even or uneven size and have <10% of the volume of embryos filled with anucleate fragments. Grade 3 embryos have anucleate fragments occupying between 10% and 50% of the volume of the embryos. Grade 4 embryos have anucleate fragments >50% of the volume of the embryos.

Evaluation of pregnancy Urine and blood hCG will be measured 14 days after embryo transfer, and positive results indicate biochemical pregnancy. If the gestational sac is observed with ultrasonography on 7weeks after transfer, clinical pregnancy will be confirmed. Ongoing pregnancy is defined by the presence of a gestational sac with fetal heartbeat after 12 weeks of gestation.

Follow-up For women not diagnosed pregnant in the initial cycle, they will be considered as a negative for outcome in our trial, and subsequently be treated another IVF/ICSI cycle or are evaluated as not suitable for further ART, based on the physician's decision.

For women who are confirmed as ongoing pregnancy, we will arrange 3 telephone interviews during their pregnancy via specific trained nurses. At 12 weeks, 28 weeks, and 37 weeks of gestation (in terms of first-trimester pregnancy, second-trimester pregnancy, and third-trimester pregnancy), pregnancy complications, and fetus information will be collected and recorded to complete the case report form (CRF) comprehensively.

Participants will be required to notify researchers of the time of delivery. In 2 weeks after delivery, the delivery information (gestational age, delivery mode, placenta abnormality and/or delivery complications), infant information (such as sex, birth weight, birth defect) will be collected by completing forms designed for this visit.

After informed consent obtained, researchers should collect the demographic characteristics, medical record, and vital signs from participants, including birth date, age, height, weight, household income and occupation for demographic characteristics; disease history, operation history and personal history for medical record; body temperature and blood pressure for vital signs.

Baseline characteristics of patient's accessory examination, such as chest radiograph, electrocardiogram (ECG), liver enzyme, renal function, HBV/HCV/HIV negative status, syphilis detection, et al.

During the study procedures, laboratory tests should be obtained to confirm the eligible criteria and collect study information, including serum sex hormone (E2, LH, FSH, PRL, P, T), ultrasonography, semen analysis, and pregnancy test. Other laboratory indexs will be tested during conventional clinical treatment but not recorded in our study.

Statistical Plans Two-Sample T-Test Power Analysis Numeric Results for Two-Sample T-Test Null Hypothesis: Mean1=Mean2. Alternative Hypothesis: Mean1<Mean2 The standard deviations were assumed to be unknown and equal. Allocation Power N1 N2 Ratio Alpha Beta Mean1 Mean2 S1 S2 0.90041 354 354 1.000 0.02500 0.09959 5.2 6.2 4.1 4.1 Report Definitions Power is the probability of rejecting a false null hypothesis. Power should be close to one.

N1 and N2 are the number of items sampled from each population. To conserve resources, they should be small.

Alpha is the probability of rejecting a true null hypothesis. It should be small.

Beta is the probability of accepting a false null hypothesis. It should be small.

Mean1 is the mean of populations 1 and 2 under the null hypothesis of equality. Mean2 is the mean of population 2 under the alternative hypothesis. The mean of population 1 is unchanged.

S1 and S2 are the population standard deviations. They represent the variability in the populations.

Summary Statements Group sample sizes of 354 and 354 achieve 90% power to detect a difference of -1.0 between the null hypothesis that both group means are 5.2 and the alternative hypothesis that the mean of group 2 is 6.2 with estimated group standard deviations of 4.1 and 4.1 and with a significance level (alpha) of 0.02500 using a one-sided two-sample t-test. Considering a 15% dropout rate in the study, 834 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 and <42 years old
* AFC: ≥5 and <20
* AMH: ≥1.1 ng/mL and <2.5 ng/mL
* BMI: ≥18.5 Kg/m2 and <29 Kg/m
* First or second ART cycle
* Regular menstrual cycles (between 22 and 35 days)
* Two ovaries present
* Planned for single or double day 3 transfer
* Infertile couples scheduled for their first IVF/ICSI cycle with fixed antagonist protocol.
* Informed consent obtained.

Exclusion Criteria:

* Women with contraindication for IVF or ICSI, such as poorly controlled type 1 or type 2 diabetes mellitus; undiagnosed liver disease or dysfunction (based on serum liver enzyme test results); renal disease or abnormal serum renal function; significant anemia; history of deep venous thrombosis, pulmonary embolus or cerebrovascular accident; uncontrolled hypertension or known symptomatic heart disease; history of (or suspected) cervical carcinoma, endometrial carcinoma or breast carcinoma; and undiagnosed vaginal bleeding.
* Previous history of poor ovarian response (<4 oocytes retrieved) with a maximal dose of OS (≥300 IU/day) or OHSS, regardless of gonadotropin dose
* Known reasons for impaired implantation (i.e. hydrosalpinx, fibroid distorting the endometrial cavity, Asherman's syndrome, thrombophilia or endometrial tuberculosis)
* Repeated miscarriages (>2 previous biochemical pregnancies or >2 spontaneous miscarriages)
* Recurrent implantation failure (>3 failed cycles with good quality embryos)
* PCOS
* Untreated thyroid disfunction
* Administration of exogenous E2, P4 or gonadotropins in the preceding menstrual cycle
* Active female smoking
* Ongoing pregnancy
* Women who have previously enrolled in the trial
* Those unable to comprehend the investigational nature of the proposed study
* either male partner or female partner has to receive donor sperm or donor eggs.
* Either male partner or female partner has to receive PGD and PGS.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile female could be enrolled.
Enrollment: 834 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
number of high-quality embryos | 4 weeks
  Whether delaying the trigger for 1～2 days will get more high-quality embryos than conventional trigger

SECONDARY OUTCOMES:
Cumulative live birth rate | 24 months
  Whether delaying the trigger for 1～2 days will get higher cumulative live birth rate

CONTACTS AND LOCATIONS:
Overall Officials: Li, Study Chair — Peking University Third Hospital
Locations (1):
- Peking Univesity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.